CLINICAL TRIAL: NCT04417153
Title: Who Benefits More? Optimising Mindfulness Based Interventions for Improved Psychological Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Collaborators: Potential project, www.potentialproject.com (Unknown); Brahm Centre, Singapore (Unknown)
Responsible Party: Principal Investigator, Julian Lim, Assistant Professor, National University of Singapore
Other Study IDs: S-19-176
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Stress, Psychological; Sleep Initiation and Maintenance Disorders
Keywords: Mindfulness; Covid; lockdown; Stress; Sleep
MeSH Terms: conditions — Stress, Psychological; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mindfulness based intervention, Non Emergency (MBI-NE): * 4 week Mindfulness foundation course face to face (MF-NE) or
  * 8 week Mindfulness Based stress reduction face to face (MBSR-NE)
  The mindfulness-based intervention consists of either four (MF) or eight (MBSR) 2-hour sessions. Participants will be provided handouts for the information covered during these talks and discussions.
  Classes are done at the Mindfulness centres providing the courses, with face to face sessions with the teacher and up to 30 participants together
  Interventions: Behavioral: Mindfulness Based Intervention
- Mindfulness based intervention, DORSCON Orange (MBI-Orange)): * 4 week Mindfulness foundation course face to face (MF-Orange) or
  * 8 week Mindfulness Based stress reduction face to face (MBSR-Orange)
  The content of these courses are the same as in the non emergency ones, and consist of four (MF) or eight (MBSR) 2-hour sessions covering various mindfulness techniques. Participants will also be provided with the same handouts for the information covered during these talks and discussions.
  Classes are done at the Mindfulness centres providing the courses, with face to face sessions with the teacher and up to 30 participants together.
  Interventions: Behavioral: Mindfulness Based Intervention
- Mindfulness based intervention, Partial lockdown (MBI-Covid): * 4 week Mindfulness foundation course online (MF-Covid) or
  * 8 week Mindfulness Based stress reduction online, partial lockdown situation (MBSR-Covid)
  The content of these courses are the same as in the non emergency ones. Participants will also be provided with the same handouts for the information covered during these talks and discussions.
  During the partial lockdown, classes can only be held online, using platform as zoom with the teacher and up to around 17 participants together.
  Interventions: Behavioral: Mindfulness Based Intervention

INTERVENTIONS:
Behavioral: Mindfulness Based Intervention — The mindfulness-based intervention consists of either four (MF) or eight (MBSR) 2-hour sessions covering various mindfulness techniques (e.g. mindfulness of breath, body and movement, senses and informal practice, and empathy and compassion). Participants will be provided handouts for the information covered during these talks and discussions.These can be done either face to face or online.
  Other Names: MBI

SUMMARY:
Mindfulness training has been gaining popularity in the past decade as a means of improving general well-being. This trend appears in response to the new stressors that have arisen with the increased stress of the 21st century. Studies have shown that the psychological state of metacognitive awareness encapsulated in mindfulness can promote the decreasing of stress as well as the secondary effect of improving sleep quality; both outcome measures of this study. While the body of research evaluating these benefits is growing, there is limited emphasis placed on the individual differences that can affect the overall efficacy of mindfulness training.

Our aim in this study is to observe the effects of mindfulness training on perceived stress levels as well as on sleep using subjective measures in a large sample of trainees. To achieve this, participants will be recruited from a pool of people who have signed up for a 4-week foundational mindfulness or 8-week mindfulness based stress reduction course at Brahm Centre. Questionnaires will be administered both before and after these courses to evaluate both stress levels and sleep habits as well as other factors which could contribute to the efficacy of mindfulness training. These inventories will probe the different facets of interpersonal differences that could serve to influence the effectiveness of the mindfulness intervention. In addition, the investigators will also test the effect of conducting the course online during a situation of emergency, like it is the partial lockdown that was implemented in Singapore due to the spread of Covid-19.

The proposed study has the potential to provide new insights into the factors that affect the efficacy of mindfulness on stress and sleep, in a situation of non-emergency (until February the 6th 2020) as well as during a period of heightened restrictions (DORSCON Orange, from 7th of February to 6th of April 2020) and a partial lockdown (from 7th of April to 1st of June 2020, or until resume of normal activity). Further, the investigators hope to build an algorithm that can predict the potential effectiveness of mindfulness on a person by person basis. This could serve as a foundation for future recommendations for mindfulness training as well as open the door for future studies that could serve to further customize the mindfulness training framework to accommodate individual differences

DETAILED DESCRIPTION:
Health and well-being are increasingly being emphasized in modern society. In response, mindfulness-based training (MBT) (e.g. Mindfulness Based Stress Reduction (MBSR) (Kabat-Zinn,1990)) is slowly gaining popularity as a method to alleviate the stress of modern day living. MBT involves bringing one's attention to the present moment, stopping one's thoughts from drifting into concerns about the past or the future It has significant effects on improving mental health via reducing symptoms of stress, anxiety and depression (Fjorback, Arendt, Ørnbøl, Fink & Walach, 2019). Local studies have similarly demonstrated the efficacy of mindful training in stress reduction for mental health professionals in Singapore (Suyi, Meredith & Khan, 2017).

Reducing stress and improving metacognitive processes also contributes to better emotional regulation, thus facilitating better sleep quality (Chiesa et al., 2011; Zeidan et al., 2010).. By breaking up cycles of rumination and worry, mindfulness is hypothesized to reduce "verbal overregulation" and facilitate the disengagement necessary to fall asleep (Gross et al., 2011). Mindfulness programs have been found to improve sleep quality in both healthy individuals (Lazar et al., 2000) and patients with medical or psychiatric illness, including insomnia and depression (Carlson & Garland, 2005; Heidenreich et al., 2006).

While there is much documentation supporting the efficacy of mindfulness training on stress and sleep, there is little research that attempts to evaluate the interpersonal differences or factors that predict the efficacy of mindfulness training on sleep and stress. Isolating these predictive variables consequently allows a better way to evaluate suitability of the mindfulness intervention on an individual basis; maximizing the results for the individual. With this new information, individuals suffering from stress and bad sleep would be able to better be able to select the most effective intervention.

While the concepts above have often been explored in relation to mindfulness, no studies to date have used machine learning to assess how these variables predispose an individual to benefit from mindfulness training. Generating this algorithm will allow for the prediction of treatment response in future trainees. Further, a better understanding of the effect of individual differences on efficacy can open the door for future research to examine how and why these differing results exist and incorporate this information to increase the effectiveness of mindfulness training.

Participants signing up for the 4 or 8 weeks mindfulness training courses at the Brahm Centre and run by Potential Project (two external organization providing Mindfulness based courses) will be automatically sent a link to the questionnaire packet several days after course enrolment. Participants will be provided with a survey link in the enrolment email that is sent to participants to confirm their enrolment, separate recruitment e-mails will not be sent out.

Participants will be informed that the data will form part of a research study, that any information provided is anonymous, and that they can opt out of completing the questionnaires without any penalty to their class enrolment. Recruitment emails will not be sent out. On enrollment in any of the courses, participants will be informed that there is an option to take part in the study.

Staff sending out emails will be separate from staff carrying out the mindfulness training programs. This will ensure that there will be no scenario where a dependent relationship will occur.

Participants can decide if they prefer to sign up for the 4 weeks or 8 weeks Mindfulness courses, depending on availability at the Mindfulness centres.

Questionnaires will be administered through the platform SurveyMonkey ©. SSL encryption will be used to protect sensitive data as it is relayed between the respondent's computer and SurveyMonkey© servers.

Questionnaires will be administered twice, with the predictor surveys administered at pre-intervention only, and outcome variables collected both pre- and post-intervention (PSQI and PSAS).

Predictive factors 10 predictive factors were chosen to evaluate their predictive qualities on the effectiveness of mindfulness training in reducing stress and improving sleep: Personality: Mindfulness training has been shown to be more effective in students with higher scores in conscientiousness and neuroticism (Winning & Boag, 2015). As such, the NEO-FFI-3 will be used to measure the dimensions of personality.

Trait Mindfulness: Baseline trait mindfulness has been shown to be a significant moderator of MBSR intervention effects (Shapiro, Brown, Thoresen, & Plante, 2010). The investigators have included trait mindfulness to corroborate previous studies that have shown this relationship as well as to explore its effect within a local population.

Mood and depression: While depression and mood has been often measured in conjunction with Mindfulness training, there has been little to no research on how it relates to mindfulness training efficacy State-Trait Anxiety: Mindfulness has been shown to alleviate state trait anxiety in individuals (Bergen-Cico & Cheon, 2013). The investigators are thus interested in whether a higher or lower baseline score in the STAI will affect the efficacy of mindfulness training Empathy: There are mixed results in regards to the relationship between empathy and mindfulness; with some studies finding no significant connection (Bergen-Cico & Cheon, 2013), and others showing differing effectiveness dependent on personality traits (Winning & Boag, 2015; Ridderinkhof, de Bruin, Brummelman, & Bögels, 2017).

Self-compassion: Self compassion is believed to be developed and enhanced through mindfulness training. Birnie, Speca & Carlson (2010) found strong associations between self-compassion and mindfulness. It was found that changes in self-compassion were predictive of changes in mindfulness.

Learning styles: This was included to investigate whether the difference in learning styles in individuals would affect the ways in which the mindfulness training are internalized; in turn influencing the efficacy of mindfulness training.

Expectancy/Credibility: Expectancy has been shown to be predictive in evaluating the outcome on some measures (Devilly & Borkovec, 2000). It would be beneficial to understand its effect on the effectiveness of mindfulness training.

Emotional Regulation: Emotion regulation has been shown to improve with mindfulness-based interventions (Guendelman, Medeiros & Rampes, 2017). The investigators are interested in understanding the effect of emotional regulation on mindfulness training.

Coping Methods: Mindfulness has been shown to affect the coping strategies used in individuals. The effect of coping methods on mindfulness training efficacy is thus of interest to our study.

Questionnaires Pittsburgh Sleep Quality Index (PSQI; Buysse et al., 1989)

Perceived Stress Scale (PSS; Cohen, Kamarck & Mermelstein,1983)

Objectives

This research has four objectives:

To corroborate findings on the effect of mindfulness training on perceived stress.

Hypothesis: based on previous literature, the investigators predict that mindfulness interventions will decrease perceived stress, with lower PSS score post intervention.

To test whether individual differences might be predictive of the effectiveness of mindfulness training on stress Hypothesis: through the use of machine learning, the investigators aim to create a model that can predict changes in perceived Stress (PSS) post intervention based on individual predictors as defined above.

To test whether individual differences might be predictive of the effectiveness of mindfulness training on sleep Hypothesis: through the use of machine learning, the investigators aim to create a model that can predict changes in Sleep quality (PSQI) post intervention based on individual predictors as defined above.

To test the effects of group mindfulness interventions on stress and sleep quality during a period of global uncertainty, a partial lockdown due to the COVID-19 pandemic, compared to Mindfulness intervention in a non-emergency situation.

Hypothesis (i):the investigator predict that participants would report higher levels of perceived stress and poorer sleep quality at baseline during the period of the pandemic (DORSCON Orange and lockdown) relative to an earlier control period; Hypothesis (ii): the investigators predict that online mindfulness training (during lockdown) would have be non-inferior/equivalent in reducing perceived stress and improving sleep quality compared with DORSCON Orange and the control period.

ELIGIBILITY:
Inclusion Criteria:

* Any individual above 21 years old enrolled in Mindfulness-Based Stress Reduction/Mindfulness Foundation course at Brahm Centre or with a mindfulness course with Potential Project can be included in the study.

Exclusion Criteria:

* no exclusion criteria

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any individual above 21 years old enrolled in Mindfulness-Based Stress Reduction/Mindfulness Foundation course at Brahm Centre or with a mindfulness course with Potential Project Singapore that is also interested in participating in the study.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-09-20 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Subjective measures of Sleep quality: Pittsburgh Sleep Quality Index total Score | Up to one month
  Pittsburgh Sleep Quality Index Score (PSQI) is a 19-item self-rated questionnaire for evaluating subjective sleep quality over the previous month. The PSQI has a sensitivity of 89.6% and specificity of 86.5% for identifying cases with sleep disorder, using a cut-off score of 5. The first 4 items are open questions, whereas items 5 to 19 are rated on a 4-point Likert scale. Individual items scores yield 7 components. A total score, ranging from 0 to 21, is obtained by adding the 7 component scores. A score above 5 suggests poor sleep quality. A decrease in PSQI score following intervention would reflect and improvement of sleep quality
Change in subjective measures of Stress: Perceived Stress Scale (PSS) | Up to one month
  The PSS measures whether different aspects of life were perceived as stressful by participants on a 5-point scale (where 0 was never and 4 was very often) in the past month. Positively worded questions are reversed scored and all 10 questions ratings are summarised into a total score, which ranges from 0 to 40, with higher scores indicating more perceived stress.

SECONDARY OUTCOMES:
Change in Subjective Time in Bed (TIB) | Up to one month
  Measured within the Pittsburgh Sleep Quality Index questionnaire. This is the total perceived time in bed in minutes, calculated as item 3 of the PSQI ("When have you usually gotten up in the morning?") minus item 1 ("When have you usually gone to bed?")
Change in Subjective Total Sleep Time (TST) | Up to one month
  Measured within the Pittsburgh Sleep Quality Index questionnaire. Total sleep time reflects the amount of time in minutes participants were effectively sleeping while in bed, without periods of wakefulness, on average over the past month. This will be measured by item 4 of the PSQI questionnaires: "How many hours of actual sleep do you get at night?".
Change in Subjective Sleep Onset Latency (SOL) | Up to one month
  Measured within the Pittsburgh Sleep Quality Index. This is the perceived time, in minutes, that takes participants to fall asleep from the moment they go to bed. This corresponds to item 2 of the PSQI: "How long (in minutes) has it taken you to fall asleep each night?"
Change in Subjective Wake After Sleep Onset (WASO) | Up to one month
  Measured within the Pittsburgh Sleep Quality Index questionnaire. In addition to Sleep Onset Latency (Secondary outcome 1), a second subjective measure of sleep quality is extracted from the PSQI: time of perceived wakefulness occurring after defined sleep onset. WASO is calculated by taking into account the total time spent in bed (TST) minus total sleep time (TST) and minus sleep onset latency (SOL), in minutes. High WASO scores reflect low sleep continuity and poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Lim, PhD, Principal Investigator — National University of Singapore
Locations (1):
- National University Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Carlson LE, Speca M, Patel KD, Goodey E. Mindfulness-based stress reduction in relation to quality of life, mood, symptoms of stress and levels of cortisol, dehydroepiandrosterone sulfate (DHEAS) and melatonin in breast and prostate cancer outpatients. Psychoneuroendocrinology. 2004 May;29(4):448-74. doi: 10.1016/s0306-4530(03)00054-4. PMID 14749092
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Fjorback LO, Arendt M, Ornbol E, Fink P, Walach H. Mindfulness-based stress reduction and mindfulness-based cognitive therapy: a systematic review of randomized controlled trials. Acta Psychiatr Scand. 2011 Aug;124(2):102-19. doi: 10.1111/j.1600-0447.2011.01704.x. Epub 2011 Apr 28. PMID 21534932
- [Background] Heidenreich T, Tuin I, Pflug B, Michal M, Michalak J. Mindfulness-based cognitive therapy for persistent insomnia: a pilot study. Psychother Psychosom. 2006;75(3):188-9. doi: 10.1159/000091778. No abstract available. PMID 16636636
- [Background] Kabat-Zinn, J. (1990) Full catastrophe living: Using the wisdom of your body and mind to face stress, pain and illness. New York: Delacourt.
- [Background] Birnie, K., Speca, M., & Carlson, L. (2010). Exploring self-compassion and empathy in the context of mindfulness-based stress reduction (MBSR). Stress And Health, 26(5), 359-371. doi: 10.1002/smi.1305
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Suyi Y, Meredith P, Khan A. Effectiveness of Mindfulness Intervention in Reducing Stress and Burnout for Mental Health Professionals in Singapore. Explore (NY). 2017 Sep-Oct;13(5):319-326. doi: 10.1016/j.explore.2017.06.001. Epub 2017 Jul 1. PMID 28780213